

# Informed Consent/Authorization for Participation in Research

Title of Research Study:

Impact of diaphragmatic breathing coaching on deep inspiration breath hold reproducibility and organ protection

Study Number:

2024-1120

Principal Investigator:

Melissa Mitchell, MD, PhD

## **Key Information**

Participant's Name

The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

Medical Record Number

# Why am I being invited to take part in a research study?

You are invited to take part in a research study because you have invasive breast cancer and your doctor has recommended radiation therapy.

# What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

# Why is this research being done?

Deep inspiratory breath hold is a technique that can help move the heart and lungs away from the radiation treatment area. The goal of this clinical research study is to learn if coaching patients on diaphragmatic breathing will help patients to take larger, more reproducible breaths and feel less anxiety about their treatments. Researchers hope to learn whether patients who undergo breathing coaching have better



reproducibility, larger lung capacity, and less anxiety than patients who do not undergo breathing coaching.

### How long will the research last and what will I need to do?

You are expected to be in this research study for the duration of your radiation treatment.

You will be asked to undergo a lung function test (called a spirometry test) about 1 week before CT simulation and at CT simulation as well as answer a questionnaire about treatment anxiety and satisfaction during these visits and at weekly standard of care visits.

More detailed information about the study procedures can be found under "What happens if I agree to be in this research?"

#### Is there any way being in this study could be bad for me?

Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. Some patients may experience anxiety with spirometry testing.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

# Will being in this study help me in any way?

It cannot be promised that there will be any benefits to you or others from your taking part in this research. However, the study intervention may help to reduce patient anxiety about radiation treatment, improve patient experience, and reduce radiation toxicity by minimizing heart and lung exposure. Future patients may benefit from what is learned.

# What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

Your alternative to participating in this research study is to not participate.



# **Detailed Information**

The following is more detailed information about this study in addition to the information listed above.

## Who can I talk to if I have questions or concerns?

If you have questions, concerns, or complaints, or think the research has hurt you, contact the research team at 713-858-9739 or mpmitchell@mdanderson.org.

This research has been reviewed and approved by the MD Anderson Institutional Review Board (IRB – an ethics committee that reviews research studies). You may talk to them at 713-792-6477 or IRB Help@mdanderson.org if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

### How many people will be in this study?

It is expected about 40 people will be enrolled in this research study.

## What happens if I agree to be in this research?

#### **Study Groups**

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups: the Standard Patient Education group or the Breathe Radiation Protocol Coaching group. This is done because no one knows if one study group is better, the same, or worse than the other group.

If you are in the Standard Patient Education group, you will receive standard of care patient education.

If you are in the Breathe Radiation Protocol Coaching group, you will have access to a video that helps guide you through a relaxed breath hold for the radiation treatment and also access to a coach for questions about the breathing process during radiation. This coaching will take place in the week before you undergo radiation planning.

### **Study Visits**

#### About 1 week before CT simulation:

You will have a lung function test (spirometry).



- This test measures the flow of your breathing and the volume of air in your lungs. You will sit upright in a chair with your legs uncrossed and feet flat on the ground. A clip will be placed on your nose, and you will be given a plastic mouthpiece connected to the spirometry machine. You will place your lips tightly around the mouthpiece and be asked to take in as big and deep a breath as possible and then blow out as hard and fast as you can.
- You will be asked to answer a questionnaire about treatment anxiety and satisfaction. This should take about 5 minutes to complete.

#### **During CT simulation:**

- You will have a lung function test (spirometry).
- You will be asked to answer a questionnaire about treatment anxiety and satisfaction. This should take about 5 minutes to complete.

#### During your weekly standard of care visits:

 You will be asked to answer a questionnaire about treatment anxiety and satisfaction. This should take about 5 minutes to complete.

All research will be done at the Mays Clinic, Department of Radiation Oncology.

Data such as your cancer stage, age, medications, BMI, smoking history, vitals, pain scores, scans, etc., will be collected from your medical record.

## What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you. You may withdraw from participation in this study without any penalty or loss of benefits. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

# Is there any way being in this study could be bad for me? (Detailed Risks)

Measurement of lung function by **spirometry** may cause temporary anxiety or lightheadedness.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.



Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

You will be told about any new information that may affect your health, welfare, or choice to stay in the research.

#### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant or breastfeed a baby while on this study. You must use birth control during the study if you are sexually active. If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away. Getting pregnant will result in your removal from this study.

# Will it cost anything to be in this study? Will I be paid to be in this study?

There will be no cost to you for participating in this study.

You and/or your insurance provider will not have to pay for certain research exams and procedures done that are covered by the study.

You and/or your insurance provider will be responsible for the costs of routine clinical services (such as diagnostic/therapeutic procedures, drugs, devices, laboratory assays, and other services that would ordinarily be ordered for medical care, regardless of whether or not you are participating in a study). There may be extra costs that are not covered by your medical plan that you will have to pay yourself.

Taking part in this study may result in added costs to you (such as transportation, parking, meals, or unpaid leave from work). You may have to visit the clinic/hospital more often than if you were not participating in this study.

If you have insurance, talk to your insurance provider and make sure that you understand what your insurance pays for and what it does not pay for if you take part in this study. Also, find out if you need approval from your plan before you can take part in the study.

You may ask that a financial counselor be made available to you to talk about the costs of this study.

You will not receive any compensation for taking part in this study.



## What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who need to review this information. Complete secrecy cannot be promised. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

Any personal information that could identify you will be removed or changed before data are shared with other researchers or results are made public.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

The sponsor, monitors, auditors, the IRB, and the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

Federal law provides additional protections of your medical records and related health information. These are described below.

# Will my data or samples be used for future research?

Your personal information is being collected as part of this study. These data and may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.



In some cases, all of your identifying information may not be removed before your data are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the MD Anderson IRB before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

If identifiers are removed from your identifiable private information that is collected during this research, that information could be used for future research studies or shared with another researcher for future research studies without your additional informed consent.

#### What else do I need to know?

MD Anderson may benefit from your participation and/or what is learned in this study.

Your information (both identifiable and de-identified) may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

# Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will do its best to protect the privacy of your records, but it is possible that once information is shared with people listed on this form, it may be released to others. If this happens, your information may no longer be protected by federal law.



D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.



#### **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performed un protocol. | nder this |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or h representative, using language that is understandable and appropriate. have fully informed this participant of the nature of this study and its post and risks and that the participant understood this explanation. | I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |